CLINICAL TRIAL: NCT05000567
Title: Relationship Between Eccentric Hamstring Strength and Passive Muscle Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B6702020000684
Record Dates: First submitted 2020-11-05; First posted 2021-08-11 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hamstring Injury
Keywords: Hamstrings; Stiffness; Strength; Shear wave elastography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No intervention.
- Experimental Older group (Experimental): 12 week strength training program: Nordic Hamstring Exercise
  Interventions: Other: 12 week nordic hamstring exercise program
- Experimental Younger group (Experimental): 12 week strength training program: Nordic Hamstring Exercise
  Interventions: Other: 12 week nordic hamstring exercise program

INTERVENTIONS:
Other: 12 week nordic hamstring exercise program — 12 weeks progressive eccentric strength training program targetting the hamstring muscles.
  Arms: Experimental Older group; Experimental Younger group

SUMMARY:
Ninety male subject will be divided into three group: a younger group (18-22y), an older group (30-40y) and a control group (18-40y). The study comprises 3 phases. PHASE 1: baseline strength and stiffness measurements of the hamstring muscles, PHASE 2: 12 week Nordic Hamstring strength training program (not for the control group) and PHASE 3: final strength and stiffness measurements. The aim of this study is twofold, namely to investigate (1) whether there is a difference in baseline stiffness of the hamstring muscle complex between different age categories and (2) the evolution of hamstring muscle stiffness during an eccentric strength training program within the different age groups. These two research questions could ultimately lead to a possible answer on the question if the higher probability of HSI (=hamstring strain injury) in the older age category with the lowest levels of eccentric hamstring strength could be due to an age-related difference in hamstring stiffness.

DETAILED DESCRIPTION:
Ninety male subjects will be equally allocated, according to their age, to either the younger NHE (Nordic Hamstring Exercise) group (aged between 18 and 22 years), the older NHE group (aged between 30 and 40 years) or the control group (aged between 18 and 40 years old). Potential candidates will be excluded from this study if they have a history of hamstring injuries, or a recent severe trauma or surgery in the lower extremity. All participants must perform at least 1 hour of weekly sport participation and do not participate in more than 3 training sessions a week. To ensure valid measurements of eccentric strength and muscle shear modulus, subjects will be instructed not to engage in strenuous training or sport activities 48 h prior to testing. All participants will be informed regarding the aim, content and possible risks associated with the experimental approach before they will be asked to sign an institutionally approved informed consent document, indicating voluntary participation in this study. Prior to the first training session, participants will undergo both a bilateral isokinetic eccentric and concentric strength protocol and an ultrasound elastographic assessment of the hamstring muscles to determine baseline strength (eccentric and concentric) and shear modulus of the posterior thigh muscles, respectively. Participants will be instructed not to engage in strenuous training or sport activities 48 h prior to testing to ensure a valid measure of the hamstring muscle-tendon elasticity. After completion of all the pre-training assessments, participants in the NHE groups will be familiarized with the correct execution-modalities of the eccentric hamstring exercise (NHE). For a period of 12 weeks, both experimental groups will perform a progressive eccentric strength training program targeting the hamstring muscles, solely consisting of the NHE. On the other hand, the control group will be instructed not to engage in any lower limb strength training. After completing the final training session, hamstring eccentric strength and shear modulus of all participants will be reassessed. The isokinetic strength protocol will be systematically conducted after all shear modulus measurements have been finished in order to avoid acute influences of previous exertion on the elasticity measurements.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 1h sport/week and Maximum 3 sport sessions a week
* Male
* Injury-free at the moment of testing.

Exclusion Criteria:

* History of injuries or surgery lower extremity
* History of hamstring injuries

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in hamstring muscle stiffness, measured by a Shear Wave elastography device. | At baseline and after 12 weeks.
  Via Shear Wave Elastography, the stiffness of the hamstring muscles (long head of the biceps femoris muscle, semitendinosus muscle and semimembranosus muscle) will be assessed. A shear wave elastography device (Aixplorer, version Mach 30, Supersonic Imagine, Aix-en-Provence, France) coupled with a linear transducer array (SL 18-5, 5-18 MHz. Super Linear, Vermon, Tours, France) will be used, in SWE mode (musculoskeletal preset, penetrate mode, smoothing level 5, persistence off, scale 0-100 kPa), to measure the shear modulus of the hamstrings (long head of the biceps femoris muscle, semitendinosus muscle and the semimembranosus muscle). The muscle stiffness will be depict by the passive shear modulus expressed in kilopascals (kPa).
  Measurement: Hamstring muscle stiffness Measurement tool: Shear wave elastography Unit of measure: Shear modulus (kPa)
Change in eccentric strength (Peak Torque) of the hamstring muscle measured by a BIODEX 4 isokinetic device. | At baseline and after 12 weeks.
  Via the BIODEX 4 isokinetic device (Biodex Medical Systems, New York, USA), the eccentric strength of the hamstring muscles will be assessed and expressed in Peak Torque (Nm/kg). The eccentric strength will be measured at two angular velocities: 30°/s and 120°/s.
  Measurement: Eccentric muscle strength of the hamstring muscles Measurement tool: BIODEX isokinetic device Unit of measure: Peak Torque (Nm/kg) at 30°/s and at 120°/s.
Change in eccentric strength (Angle of peak torque) of the hamstring muscle, measured by a BIODEX 4 isokinetic device. | At baseline and after 12 weeks.
  Via the BIODEX 4 isokinetic device (Biodex Medical Systems, New York, USA), the eccentric strength of the hamstring muscles will be assessed and expressed in Angle of Peak Torque (°). The eccentric strength will be measured at two angular velocities: 30°/s and 120°/s.
  Measurement: Eccentric muscle strength of the hamstring muscles Measurement tool: BIODEX isokinetic device Unit of measure: Angle of Peak Torque (°) at 30°/s and at 120°/s.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Principal Investigator — Departement of Rehabilitation Sciences, Ghent University
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No